CLINICAL TRIAL: NCT03013907
Title: Emotional Awareness and SElf-regulation for Depression in Patients With Hypertension (EASE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01350
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hypertension
Keywords: Hypertension; Coping; Relaxing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPLIFT (Experimental): Eligible participants will complete 8 weekly group sessions by phone. The intervention builds cognitive-behavioral and mindfulness skills to help reduce depressive symptoms. Each hour-long weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.
  Interventions: Behavioral: UPLIFT
- Usual Care (Active Comparator): Subjects randomized to UC will be advised to seek help from their primary care physician (PCP) or other sources as they normally would if they encountered symptomatic deterioration or other difficulties over the course of the study. All treatments received over the course of the study for the UC group and outside of the study (for the intervention group) will be assessed at each time point.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: UPLIFT — Session 1: Introduction to UPLIFT/Noticing Thoughts Session 2: Checking and Changing Thoughts Session 3: Coping & Relaxing Session 4: Attention & Mindfulness Session 5: The Present as a Calm Place Session 6: Thoughts as Changeable, Thoughts as Not Fixed Session 7: Focus on Pleasure & the Importance of Reinforcement Session 8: Preventing Lapses and Giving Thanks
  Arms: UPLIFT
Behavioral: Usual care — Subjects randomized to UC will be advised to seek help from their primary care physician (PCP) or other sources as they normally would if they encountered symptomatic deterioration or other difficulties over the course of the study
  Arms: Usual Care

SUMMARY:
The purpose of this study is to adapt and then evaluate the feasibility, acceptability, and efficacy of a telephone-based intervention (UPLIFT: Using Practice and Learning to Increase Favorable Thoughts) for individuals with elevated depressive symptoms and hypertension. UPLIFT is a group-based intervention that is delivered over 8 weekly sessions for 1 hour/week by phone.

Aim 1 of this study is to adapt UPLIFT using qualitative focus groups and individual interviews and to test the adapted UPLIFT program in a single-arm design. Aim 2 of this study is a randomized controlled trial (RCT) that will compare the effects of the adapted UPLIFT program to usual care (UC) and to test mediators and moderators of the effects of UPLIFT.

DETAILED DESCRIPTION:
Once 16 participants are enrolled (to form 2 groups of 8 patients each), an independent study staff member will determine participants' group assignments. The randomization sequence will be created a priori by Dr. Keith Goldfeld (biostatistician) by using a computer-generated list of random numbers with stratification by antidepressant medication use and baseline levels of depressive symptoms (PHQ scores <10 and ≥10).

UPLIFT: Eligible participants will complete 8 weekly group sessions by phone. The intervention builds cognitive-behavioral and mindfulness skills to help reduce depressive symptoms. Each hour-long weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.

Usual care: Subjects randomized to UC will be advised to seek help from their primary care physician (PCP) or other sources as they normally would if they encountered symptomatic deterioration or other difficulties over the course of the study. All treatments received over the course of the study for the UC group and outside of the study (for the intervention group) will be assessed at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension based on the criteria in the ICD-9/-10
* Mild to moderate depressive symptoms (PHQ-9 ≥ 5)
* English-speaking
* If taking depression medications, medications must stable for the past 6 weeks (no change to type or dose)
* Willing to provide informed consent, be audio-recorded, and comply with all other aspects of protocol

Exclusion Criteria:

* Moderate to severe depressive symptoms (PHQ-9 ≥ 15)
* Current substance abuse
* Current eating disorder
* Self-harm within the past 3 months
* Current obsessive-compulsive disorder
* Current anxiety disorder (e.g., PTSD, panic disorder)
* Active suicidal ideation
* History of or current diagnosis of psychosis
* Significant cognitive impairment (mini mental state examination score ≤ 20)
* History of previous training in mindfulness
* History of more than 8 sessions of cognitive behavioral therapy
* Counseling more frequently than once per month

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by the number of weekly sessions attended | 6 Months
  Determined by the number of weekly sessions attended and number of days of home-based practice completed each week
Acceptability | 6 Months
  8-item Client Satisfaction Questionnaire (CSQ-8)
PHQ-9 | 6 Months
  validated measure of depressive symptoms. Items rate symptom severity during the prior 2 weeks based on DSM-IV diagnostic criteria for major depression. Scores range from 0-27; scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively. The PHQ-9 will be completed at screening and at all study visits (continuous scores).
Quick Inventory of Depressive Symptomatology (QIDS-SR 16) | 6 Months
  Standardized depression instrument that has treatment sensitivity advantages over the PHQ-9 and will be administered at pre- and post-treatment. Total scores on the QIDS-SR16 range from 0 to 27 and reflect depression severity across 9 domains of the DSM-IV MDD criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Shallcross, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States